CLINICAL TRIAL: NCT07358390
Title: Potatoes as a Strategy to Improve Diet Quality in Young Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Emily Hohman, Associate Research Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00027376
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dietary Intake
Keywords: vegetables; potatoes; preschool; Head Start
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Intervention Model Description: Participants will complete four conditions in a randomized order.
Masking Description: The intervention consists of different combinations of potatoes and vegetables, and data collection includes food intake, and thus masking is not possible for participants or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Randomization order 1 (Experimental): Participants will complete the four conditions in the following order: 1) potato + vegetable, 2) potato appetizer, 3) no potato, and 4) potato and vegetable separate
  Interventions: Other: Potato + vegetable; Other: Potato appetizer; Other: Potato and vegetable separate; Other: No potato
- Randomization order 2 (Experimental): Participants will complete the four conditions in the following order: 1) no potato, 2) potato + vegetable, 3) potato and vegetable separate, and 4) potato appetizer
  Interventions: Other: Potato + vegetable; Other: Potato appetizer; Other: Potato and vegetable separate; Other: No potato
- Randomization order 3 (Experimental): Participants will complete the four conditions in the following order: 1) potato and vegetable separate, 2) potato appetizer, 3) no potato, and 4) potato + vegetable
  Interventions: Other: Potato + vegetable; Other: Potato appetizer; Other: Potato and vegetable separate; Other: No potato
- Randomization order 4 (Experimental): Participants will complete the four conditions in the following order: 1) potato appetizer, 2) no potato, 3) potato and vegetable separate, and 4) potato + vegetable
  Interventions: Other: Potato + vegetable; Other: Potato appetizer; Other: Potato and vegetable separate; Other: No potato
- Randomization order 5 (Experimental): Participants will complete the four conditions in the following order: 1) no potato, 2) potato and vegetable separate, 3) potato + vegetable, and 4) potato appetizer
  Interventions: Other: Potato + vegetable; Other: Potato appetizer; Other: Potato and vegetable separate; Other: No potato
- Randomization order 6 (Experimental): Participants will complete the four conditions in the following order: 1) potato + vegetable, 2) potato and vegetable separate, 3) potato appetizer, and 4) no potato
  Interventions: Other: Potato + vegetable; Other: Potato appetizer; Other: Potato and vegetable separate; Other: No potato

INTERVENTIONS:
Other: Potato + vegetable — A mixed dish of potatoes and other vegetables will be served at lunch
Other: Potato appetizer — A potato dish will be served as an appetizer at lunch prior to the main course
Other: Potato and vegetable separate — A potato dish and a vegetable dish will be served separately at lunch
Other: No potato — No potato dish will be served at lunch

SUMMARY:
The purpose of this study is to examine whether incorporating potatoes into meals-either paired with other vegetables or served as a first course-can improve preschoolers' vegetable intake, reduce excess energy intake, and improve overall diet quality. Findings will be used to inform whether potatoes, a well-liked and commonly consumed vegetable, could be leveraged in several ways to improve the overall diet quality of children.

DETAILED DESCRIPTION:
The overall object of this study is to test potato-based strategies to improve diet quality in preschool age children. The specific aims are:

Aim 1: Determine if pairing potatoes with other less-preferred vegetables increases liking and intake of the non-potato vegetables.

Aim 2: Determine if potato-based dishes can be used strategically to reduce intake of more energy-dense entrees.

The effect of potato-based dishes on vegetable intake and total energy intake will be tested across four lunch-time sessions in preschool classrooms. Each lunch session will be randomly assigned to one of the potato dish conditions.

ELIGIBILITY:
Inclusion Criteria:

Child:

* Enrolled in participating Head Start classroom
* Age 2-6 years old

Parent:

* Parent/guardian of a participating child
* Age 18 years or older
* Able to read and answer questions in English

Teacher:

* Teacher/teaching staff member of a participating Head State classroom
* Age 18 years or older
* Able to read and answer questions in English

Exclusion Criteria:

Child:

* Allergy to potatoes
* Children who are not able to understand and answer questions in English may participate in all parts of the study except for the taste test ratings, which require the child to communicate with the research assistant

Parent:

- Child not enrolled in the study

Teacher exclusion criteria:

- None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intake of target vegetable at lunch | At each of four lunch sessions conducted once per week over four weeks
  Intake of the non-potato target vegetable will be measured at each lunch session by weighing the food dish prior to serving and after the participant has finished eating
Entree intake at lunch | At each of four lunch sessions conducted once per week over four weeks
  Intake of an energy-dense entree (macaroni and cheese) will be measured at each lunch session by weighing the food dish prior to serving and after the participant has finished eating
Liking of vegetable + potato dishes | Once at start of study
  Children will be presented with small samples of several vegetable, potato, and vegetable + potato dishes and asked to taste them. Children will rate each food as 'yummy', 'just ok', or 'yucky' using a pictorial scale. We will compare the percentage of children who rate the vegetable with potato (VEG+POT) dishes as yummy to the percentage that rated the same non-potato vegetable alone (VEG) as 'yummy'.

SECONDARY OUTCOMES:
Willingness to taste vegetable + potato dishes | Once at beginning of study
  Children will be presented with small samples of several vegetable, potato, and vegetable + potato dishes and asked to taste them. Children will rate each food as 'yummy', 'just ok', or 'yucky' using a pictorial scale. We will compare the percentage of children who were willing to taste the vegetable with potato (VEG+POT) dishes to the percentage that were willing to taste the same non-potato vegetable alone (VEG).
Intake of potatoes at lunch | At each of four lunch sessions conducted once per week over four weeks
  Intake of the potato dish will be measured at each lunch session by weighing the food dish prior to serving and after the participant has finished eating
Total vegetable intake at lunch | At each of four lunch sessions conducted once per week over four weeks
  Total intake of potato and non-potato vegetables will be measured at each lunch session by weighing the food dishes prior to serving and after the participant has finished eating
Total energy intake at lunch | At each of four lunch sessions conducted once per week over four weeks
  Total energy intake in kcal will be measured at each lunch session by weighing the food dishes prior to serving and after the participant has finished eating

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Hohman, PhD, Principal Investigator — Penn State University

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared by depositing the data set and relevant metadata into a scientific data repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared after publication of the primary outcome manuscripts and will be available indefinitely.
Access Criteria: Researcher will be able to access the deidentified IPD using protocols established by the data repository.